CLINICAL TRIAL: NCT01008878
Title: Treatment of the Metabolic Syndrome in an Interdisciplinary Obesity Clinic: a Randomized Controlled Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Dr Marie-France Langlois, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 04-003
Record Dates: First submitted 2009-11-05; First posted 2009-11-06 (Estimated); Last update posted 2009-11-06 (Estimated); Status verified 2009-11

CONDITIONS: Obesity; Metabolic Syndrome
MeSH Terms: conditions — Obesity; Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: interdisciplinary intervention

SUMMARY:
This study is a randomized, controlled and opened trial designed to compare the effects of an interdisciplinary moderate-intensity lifestyle modification program vs. conventional treatment by primary care physicians.

We want to show the benefits of coherent interdisciplinary care in the obesity clinic of CHUS (Centre Hospitalier Universitaire de Sherbrooke) in comparison to the conventional treatment in order to:

* Improve subjects' characteristic features of metabolic syndrome: weight, waist circumference, fatty mass, plasma lipid profile, blood pressure, fasting glycaemia, and HbA1c;
* Improve our patients' nutritive practices;
* Decrease our patients' sedentary lifestyle;
* Improve our patients' motivation to lose weight, and to improve their quality of life; We also wish to define predictors of answer in order to better select the patients if necessary, and evaluate the costs incurred by the health system.

DETAILED DESCRIPTION:
Eligible participants recruited from patients, referred through the obesity clinic were separated into two groups.

The interdisciplinary treatment group received interventions at our clinic for 6 months.. The intervention included a visit every 6 weeks including a nursing consultation (listening, psychological support, anthropometric measurements and blood pressure), an endocrinologist consultation, a nutritionist consultation (initial evaluation of food intake and counselling), a psychologist consultation if needed, an interactive group information session (to discuss the following: diet, psychological aspects associated with obesity, physical education, complications and pharmacological treatments of obesity), and a questionnaire on the individual costs of their visit.

A control group was monitored during this 6 months by their family physician, as per usual.

A biological assessment, questionnaires, and tests will be carried out in beginning and end of program: the questionnaires are to evaluate the physical activity (Sallis, Canada fitness survey); the quality of life (IWQOL-Lite, SF-36); the motivation (analogical visual Scales); knowledge (pretest and post-test); and costs. Tests to assess physical activity (6-minute walk test and accelerometer) will also be administered.

After the first 6 months, both groups were followed at the obesity clinic for another 12 months.

ELIGIBILITY:
Criteria Inclusion:

* referred to the obesity clinic by a medical doctor;
* BMI > 27 kg/m²; (Body Mass Index)
* metabolic associated syndrome according to the definition of the NCEP-ATP III
* be able to give an inform consent

Criteria Exclusion:

* Impossibility to be present at the visits
* Physical/motor incapacity (or other) making one unable and insecure to walk at a moderate to rapid speed for 6 min and more
* Use of an anti-obesity treatment the last 3 months
* Bariatric Surgery in the past
* Planned Pregnancy
* Pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2004-03; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
After 6 months of follow-up, the treatment group proportion achieved a 5% reduction in body weight compared to the control group. | 6 months

SECONDARY OUTCOMES:
Weight; fatty mass; features of the metabolic syndrome; food intake; energy expenditure; quality of life; motivation; cost/effectiveness.
Metabolic syndrome characteristics | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Marie-France Langlois, MD, Principal Investigator — Medecine Department, Division of endocrinology, CHUS
Locations (1):
- Centre de Recherche Clinique (CRC), Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec, Canada